CLINICAL TRIAL: NCT05245500
Title: A Phase 1 Multiple Expansion Cohort Trial of MRTX1719 in Patients With Advanced Solid Tumors With Homozygous MTAP Deletion
Brief Title: Phase 1 Study of MRTX1719 in Solid Tumors With MTAP Deletion
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA240-0007; CA240-0007 (Other: Bristol-Myers Squibb Protocol ID); 1719-001 (Other: Mirati Therapeutics Protocol ID); NCT06937970 (obsolete NCT alias)
Record Dates: First submitted 2022-02-01; First posted 2022-02-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Mesothelioma; Non Small Cell Lung Cancer; Malignant Peripheral Nerve Sheath Tumors; Solid Tumor; Pancreatic Adenocarcinoma; Advanced Solid Tumor
Keywords: MTAP Deletion; Mesothelioma; Non Small Cell Lung Cancer; Malignant Peripheral Nerve Sheath Tumors; Solid Tumor; MTAP; Malignant; Pancreatic adenocarcinoma; Pancreas Cancer; PRMT5; Synthetic Lethality; Advanced Solid Tumor; NSCLC
MeSH Terms: conditions — Mesothelioma; Carcinoma, Non-Small-Cell Lung; Neurofibrosarcoma; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1/1B (Experimental): Dose Escalation/Evaluation
  Interventions: Drug: MRTX1719
- Phase 1b Sub-studies 1-4 (Experimental)
  Interventions: Drug: MRTX1719
- Phase 1b Sub-study 5 (Experimental)
  Interventions: Drug: MRTX1719

INTERVENTIONS:
Drug: MRTX1719 — MRTX1719 is a potent PRMT5-MTA inhibitor. Specified dose on specified days

SUMMARY:
This is a Phase 1, open-label, multicenter, study of the safety, tolerability, PK, PD, and anti-tumor activity of MRTX1719 patients with advanced, unresectable or metastatic solid tumor malignancy with homozygous deletion of the MTAP gene.

DETAILED DESCRIPTION:
This first-in-human clinical trial will begin with an exploration of MRTX1719 dose and regimen. As potentially viable regimens are identified, Phase 1b expansion cohorts may be implemented to ensure sufficient safety experience, PK information, compare food effect and relative bioavailability between capsules and tablets, and early evidence of clinical activity are available.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed diagnosis of a solid tumor malignancy with homozygous deletion of the MTAP gene detected in tumor tissue.
* Unresectable or metastatic disease.
* Presence of a tumor lesion amenable to mandatory biopsy for pharmacodynamic evaluation at baseline and on-study unless Sponsor-confirmed as medically unsafe or infeasible.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function.

Exclusion Criteria

* Prior treatment with a PRMT5 or MAT2A inhibitor therapy.
* Active brain metastases or carcinomatous meningitis.
* History of significant hemoptysis or hemorrhage within 4 weeks of the first dose of study treatment.
* Major surgery within 4 weeks of first dose of study treatment.
* History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions (eg, uncontrolled nausea, vomiting, malabsorption syndrome) likely to alter absorption of study treatment or result in inability to swallow oral medications.
* Cardiac abnormalities.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2027-12-10 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Number of Patients who Experience Dose-Limiting Toxicity | 21 days
Number of patients who experience a treatment-related adverse event | Up to 2 years
Objective response rate (ORR) | 2 years
Duration of response (DOR) | 2 years
Progression free survival (PFS) | 2 years
Overall survival (OS) | 2 years
Number of Patients With Clinically Significant Laboratory Assessments | Up to 4 years

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Up to 4 days
Time to achieve maximal plasma concentration (Tmax) | Up to 4 days
Maximum observed plasma concentration (Cmax) | Up to 4 days
Terminal elimination half-life (t1/2) | Up to 4 days
Apparent total plasma clearance when dosed orally (CL/F) | Up to 4 days
Apparent volume of distribution when dosed orally (Vz/F) | Up to 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- United States (24):
  - Mayo Clinic, Phoenix, Arizona
  - Sarah Cannon Research Institute (SCRI) - HealthONE Location, Denver, Colorado
  - Rocky Mountain Cancer Centers, LLP - Oncology, Lone Tree, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Orlando, Florida
  - Local Institution - 124, Chicago, Illinois
  - Dana-Farber Cancer Institute, Brookline, Massachusetts
  - Cancer and Hematology Centers of Western Michigan, Norton Shores, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Local Institution - 129, Mineola, New York
  - David H Koch, Memorial Sloan Kettering Cancer Center, New York, New York
  - New york cancer and blood specialists - Oncology, Port Jefferson Station, New York
  - University of North Carolina - Gastroenterology and Hepatology, Chapel Hill, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - Ut Southwestern, Dallas, Texas
  - Texas Oncology - DFW, Fort Worth, Texas
  - MDACC, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - Texas Oncology, P.A. - Oncology, Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Local Institution - 134, Seattle, Washington
  - Local Institution - 108, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05245500.html